CLINICAL TRIAL: NCT05864274
Title: Using a Novel Mobile Cognitive Training Application to Improve Cancer-related Cognitive Impairment in Gynecologic Oncology Patients
Brief Title: Improve Cancer-related Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Teresa Boitano, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300010880
Record Dates: First submitted 2023-04-11; First posted 2023-05-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Gynecologic Cancer; Chemotherapy Effect; Chemo-brain; Cancer-related Cognitive Difficulties
Keywords: CHEMOTHERAPY SIDE EFFECTS; GYNECOLOGIC CANCERS; CHEMO-BRAIN; CANCER-RELATED COGNITIVE IMPAIRMENT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- OBSERVATION (No Intervention): PATIENTS WILL PARTICIPATE IN THE NEUROPSYCHOLOGY EVALUATION BUT WILL NOT USE THE COGNITIVE MOBILE TRAINING APPLICATION.
- MOBILE COGNITIVE TRAINING APP (Experimental): These patients will undergo neuropsychology evaluation and use the cognitive mobile training application
  Interventions: Device: Cognitive training application

INTERVENTIONS:
Device: Cognitive training application — Patients will participate with a cognitive training application and undergo neurocognitive testing during and after chemotherapy.
  Other Names: study
  Arms: MOBILE COGNITIVE TRAINING APP

SUMMARY:
Cancer-related cognitive impairment (CRCI), also known as "chemobrain," is the cognitive decline that negatively impacts the majority of cancer patients undergoing chemotherapy, radiation, and/or hormonal treatments. This application focuses on evaluating if using a cognitive mobile training application can decrease the impact of CRCI in gynecologic oncology patients through a multidisciplinary approach with patients undergoing assessments by our neurocognitive team.

DETAILED DESCRIPTION:
Cancer-related cognitive impairment (CRCI), also known as "chemobrain," is the cognitive decline that negatively impacts the majority of cancer patients undergoing chemotherapy, radiation, and/or hormonal treatments [1]. Occurring in the majority of patients receiving cancer therapy, CRCI adverse events can, unfortunately, be lifelong and significantly affect patients' quality of life [2-4]. Given the increased lifespan of gynecologic oncology cancer patients due to the use of modern therapeutics, increased focus has been placed on evaluating quality of life during and after treatments. CRCI, alternatively known as "chemo brain" or "chemo fog" is a common side effect of cancer therapy. These symptoms frequently include augmentation of clear thinking with memory difficulties that can are very distressing to patients both during treatment and beyond. Despite effecting the majority of cancer patients, CRCI data and research is underrepresented in the gynecologic oncology population. In breast cancer, up to 77% of patient with breast cancer who received chemotherapy reported cognitive symptoms associated with the therapy [9]. In a meta-analysis looking at patient with breast cancer who were treated with chemotherapy, the most effected domains were processing speed and language, executive function, and memory [10]. In general, a significant knowledge gap in gynecologic oncology related CRCI exists as interventions to help improve this frequent and life altering group of side effects have not been evaluated to date. Therefore, to our knowledge, this proposal is the first of its kind in gynecologic oncology patients undergoing cancer therapy.

In the dementia literature, mobile applications have been utilized in cognitive training management to improve outcomes in patients [11-13]. Cognitive impairment (CI) is a precursor to dementia and can be defined as mild and major. Mild CI does not yet interfere with instrumental activities of daily living (IADLs) whereas major CI does [14]. In a recent systematic review looking at interventions to delay age-related cognitive decline, it was found that cognitive training and physical activity showed the most promise [15]. One cognitive training application (CTA) showed improvement in cognitive ability following five, fifteen-minute training applications a week for ten weeks [12]. Furthermore, a Cochrane review showed that in a group of randomized non-pharmacologic interventions in women with breast cancer, the use of cognitive training applications may reduce the risk of CRCI [16]. Unfortunately, no data currently exists on CTA use in gynecologic oncology patients. The goal of this study is to evaluate the use of a CTA in gynecologic oncology patients undergoing primary chemotherapy in order to reduce the impact of CRCI.

ELIGIBILITY:
Inclusion criteria are:

* newly diagnosed gynecologic malignancy (uterine, cervical, ovarian, primary peritoneal, vulvar, or vaginal) and undergoing chemotherapy
* own a smartphone or tablet with ability to download cognitive training application
* and age >21 years old

Exclusion criteria include:

* medical diagnosis of dementia
* significant underlying mental diagnoses for which they are on more than 1 medication for (patients with depression or anxiety on single-agent therapy will be able to participate
* age <21

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals with gynecologic cancers
Enrollment: 64 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive function | From initiation of chemotherapy through 2 years
  Evaluated by the NIH Toolbox of Assessment of Neurologic Behavioral Function
Neurocognitive function | From initiation of chemotherapy through 2 years
  Evaluated by the FACT-Cog survey

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No